CLINICAL TRIAL: NCT06195059
Title: Assessment of Pulmonary Blood Volume Using Contrast Echocardiography During Exercise
Brief Title: Contrast Echocardiography During Exercise to Assess Pulmonary Blood Volume
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Barry Borlaug, Principal Investigator, Mayo Clinic
Other Study IDs: 23-009478
Record Dates: First submitted 2023-12-19; First posted 2024-01-08 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure; Pulmonary Vascular Disease
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to evaluate whether pulmonary blood volume (PBV) derived from contrast echocardiography can serve as a non-invasive surrogate for invasive pulmonary artery wedge pressure (PAWP) during exercise. Also, to compare changes in PBV with exercise in patients with and without heart failure and pulmonary vascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the cardiac catheterization laboratory for invasive exercise right heart catheterization for evaluating exertional dyspnea. Investigators will include patients with normal or low EF, and across the spectrum of pulmonary hypertension severity.

Exclusion Criteria:

* Patient inability or unwillingness to undergo echocardiography including a contrast method, or if echocardiography would, in the opinion of the investigator, somehow compromise the quality of data acquisition for the clinical case.
* Prior adverse reaction to echo contrast administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have already been referred to the catheterization laboratory at Mayo Clinic in Rochester, MN for the exercise hemodynamic assessment will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Vascular Capacitance at Rest | Baseline
  Capacitance is defined as the total volume of blood in an organ or region at a given pressure. Pulmonary Vascular Capacitance (ml/mmHg) will be determined by pulmonary blood volume/mean pulmonary artery pressure as measured with high fidelity micromanometer catheters in the pulmonary vasculature at rest during the standard of care exercise hemodynamic assessment.
Pulmonary Vascular Capacitance During Exercise | Baseline
  Capacitance is defined as the total volume of blood in an organ or region at a given pressure. Pulmonary Vascular Capacitance (ml/mmHg) will be determined by pulmonary blood volume/mean pulmonary artery pressure as measured with high fidelity micromanometer catheters in the pulmonary vasculature during the exercise portion of the standard of care exercise hemodynamic assessment.

SECONDARY OUTCOMES:
Pulmonary Blood Volume at Rest | Baseline
  Pulmonary blood volume (ml) is measured by measuring indicator dilution curves using sonographic contrast at rest during the standard of care exercise hemodynamic assessment.
Pulmonary Blood Volume During Exercise | Baseline
  Pulmonary blood volume (ml) is measured by measuring indicator dilution curves using sonographic contrast during the exercise portion of the standard of care exercise hemodynamic assessment.
Pulmonary Vascular Compliance at Rest | Baseline
  Compliance is the change in volume for a given change in pressure. Pulmonary Vascular Compliance (ml/mmHg) is defined as stroke volume divided by Pulmonary Artery (PA) pulse pressure and will be measured with high fidelity micromanometer catheters in the pulmonary vasculature at rest during the standard of care exercise hemodynamic assessment.
Pulmonary Vascular Compliance During Exercise | Baseline
  Compliance is the change in volume for a given change in pressure. Pulmonary Vascular Compliance (ml/mmHg) is defined as stroke volume divided by Pulmonary Artery (PA) pulse pressure and will be measured with high fidelity micromanometer catheters in the pulmonary vasculature during the exercise portion of the standard of care exercise hemodynamic assessment.
Right Atrial Pressure at Rest | Baseline
  Right Atrial Pressure (mmHg) is a measure of cardiac filling pressure, measured with high fidelity micromanometer catheters in the pulmonary vasculature at rest during the standard of care exercise hemodynamic assessment.
Right Atrial Pressure During Exercise | Baseline
  Right Atrial Pressure (mmHg) is a measure of cardiac filling pressure, measured with high fidelity micromanometer catheters in the pulmonary vasculature during the exercise portion of the standard of care exercise hemodynamic assessment.
Right Ventricular Pressure at Rest | Baseline
  Right Ventricular Pressure (mmHg) is a measure of cardiac filling pressure, measured with high fidelity micromanometer catheters in the pulmonary vasculature at rest during the standard of care exercise hemodynamic assessment.
Right Ventricular Pressure During Exercise | Baseline
  Right Ventricular Pressure (mmHg) is a measure of cardiac filling pressure, measured with high fidelity micromanometer catheters in the pulmonary vasculature during the exercise portion of the standard of care exercise hemodynamic assessment.
Pulmonary Artery Pressure at Rest | Baseline
  Pulmonary Artery Pressure (mmHg) is a measure of cardiac filling pressure, measured with high fidelity micromanometer catheters in the pulmonary vasculature at rest during the standard of care exercise hemodynamic assessment.
Pulmonary Artery Pressure During Exercise | Baseline
  Pulmonary Artery Pressure (mmHg) is a measure of cardiac filling pressure, measured with high fidelity micromanometer catheters in the pulmonary vasculature during the exercise portion of the standard of care exercise hemodynamic assessment.
Pulmonary Capillary Wedge Pressure at Rest | Baseline
  Pulmonary capillary wedge pressure (mmHg) is a measure of cardiac filling pressure, measured with high fidelity micromanometer catheters in the pulmonary vasculature at rest during the standard of care exercise hemodynamic assessment.
Pulmonary Capillary Wedge Pressure During Exercise | Baseline
  Pulmonary capillary wedge pressure (mmHg) is a measure of cardiac filling pressure, measured with high fidelity micromanometer catheters in the pulmonary vasculature during the exercise portion of the standard of care exercise hemodynamic assessment.
Cardiac Output at Rest | Baseline
  Cardiac output (L/min) is the total volume of blood moved by the heart per minute and will be measured with high fidelity micromanometer catheters in the pulmonary vasculature at rest during the standard of care exercise hemodynamic assessment.
Cardiac Output During Exercise | Baseline
  Cardiac output (L/min) is the total volume of blood moved by the heart per minute and will be measured with high fidelity micromanometer catheters in the pulmonary vasculature during the exercise portion of the standard of care exercise hemodynamic assessment.
Pulmonary Vascular Resistance at Rest | Baseline
  Pulmonary vascular resistance (PVR) is the resistance against blood flow from the pulmonary artery to the left atrium. PVR (in Wood units) will be measured with high fidelity micromanometer catheters in the pulmonary vasculature at rest during the standard of care exercise hemodynamic assessment.
Pulmonary Vascular Resistance During Exercise | Baseline
  Pulmonary vascular resistance (PVR) is the resistance against blood flow from the pulmonary artery to the left atrium. PVR (in Wood units) will be measured with high fidelity micromanometer catheters in the pulmonary vasculature during the exercise portion of the standard of care exercise hemodynamic assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Borlaug, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No